CLINICAL TRIAL: NCT01041352
Title: Laryngeal Mask or Endotracheal Tube for Back Surgery in the Prone Position. Advantages, Adverse Effects and Time Consumation for the Two Methods.
Brief Title: Laryngeal Mask or Endotracheal Tube for Back Surgery in the Prone Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Karsten Skovgaard Olsen, Consultant, DMSC, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Laryngeal mask or endotracheal
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Anaesthesia; Adverse Effects
Keywords: anaesthesia; laryngeal mask; prone position
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endotracheal group (Active Comparator): airway management: endotracheal tube
  Interventions: Device: endotracheal tube
- laryngeal mask group (Active Comparator): airway management: laryngeal mask
  Interventions: Device: laryngeal mask

INTERVENTIONS:
Device: laryngeal mask — LMA Proseal
  Arms: laryngeal mask group
Device: endotracheal tube — Unomedical endotracheal tube
  Arms: Endotracheal group

SUMMARY:
The aim of the study is to compare anaesthesia (for back surgery) using endotracheal intubation (patients anaesthized in the supine position)with anaesthesia using a laryngeal mask (anaesthesia induced and the laryngeal mask placed with the patient in the prone position on the operation table) as regards advantages, adverse effects and time spent. The anaesthesia in the 2 groups of patients is identical (propofol, remifentanil, rocuronium). Two groups of 70 pt. each are included in the stud. The inclusion criterias are patients 18-70 yrs., ASA group 1-2, normal airways, patients scheduled for back surgery with an estimated duration of less than 2 hours.

Adverse effects (related to the placement on the operation table i.e. pain in the arms or shoulders, pain in the throat, blood in the sputum, irritation in the eyes etc.) and time spent with all the procedures (anaesthesia, placement of the airway, surgery and emergence from the anaesthesia are registered. The hypothesis is that the method using the laryngeal mask is faster and with fewer adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for backsurgery of an espected duration less than 2 hours,
* Age 18-70 years,
* ASA (american society of anaaesthesiology) class 1-2,
* Normal airways

Exclusion Criteria:

* Body mass index >35
* Expected time of surgery > 2 hours

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2009-10; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
time of anaesthesia | 2 years

SECONDARY OUTCOMES:
adverse effects using the 2 methods | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Karsten S Olsen, MD, DMSc, Study Chair
Locations (1):
- Glostrup University Hospital, Glostrup Municipality, Denmark

REFERENCES:
- [Derived] Olsen KS, Petersen JT, Pedersen NA, Rovsing L. Self-positioning followed by induction of anaesthesia and insertion of a laryngeal mask airway versus endotracheal intubation and subsequent positioning for spinal surgery in the prone position: a randomised clinical trial. Eur J Anaesthesiol. 2014 May;31(5):259-65. doi: 10.1097/EJA.0000000000000004. PMID 24247413